CLINICAL TRIAL: NCT04727190
Title: The Efficacy and Safety of Transbronchial Cryobiopsy vs Forceps Biopsy in the Diagnosis of Lung Ground-glass Opacity: A Prospective, Randomized Controlled Trial
Brief Title: The Efficacy and Safety of TBCB vs TBFB in Diagnosis of GGO
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Shanghai Chest Hospital (Other)
Collaborators: First Affiliated Hospital of Chongqing Medical University (Other)
Responsible Party: Principal Investigator, Jiayuan Sun, Director, Department of Respiratory Endoscopy, Shanghai Chest Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: SHCHE201904
Record Dates: First submitted 2020-03-15; First posted 2021-01-27 (Actual); Last update posted 2021-02-02 (Actual); Status verified 2021-01

CONDITIONS: Lung Ground-Glass Opacity
Keywords: Lung Ground-Glass Opacity; Transbronchial Cryobiopsy; Forceps Biopsy; Diagnosis
MeSH Terms: conditions — Disease

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TBCB group (Experimental): Specimens were obtained using 1.1 mm ultrathin cryoprobe with or without guide sheath by bronchoscope.
  Interventions: Procedure: Transbronchial Cryobiopsy
- TBFB group (Active Comparator): Specimens were obtained using 1.5 mm or 1.9 mm biopsy forceps with or without guide sheath by bronchoscope.
  Interventions: Procedure: Transbronchial Forceps Biopsy

INTERVENTIONS:
Procedure: Transbronchial Cryobiopsy — The eligible patient will be randomized to TBCB group to receive transbronchial cryobiopsy.
  Arms: TBCB group
Procedure: Transbronchial Forceps Biopsy — The eligible patient will be randomized to TBFB group to receive transbronchial forceps biopsy.
  Arms: TBFB group

SUMMARY:
The aim of this study is to investigate the difference of efficacy and safety between transbronchial cryobiopsy (TBCB) and transbronchial forceps biopsy (TBFB) in the diagnosis of lung ground-glass opacity.

DETAILED DESCRIPTION:
The conventional biopsy method for lung ground-glass opacity (GGO) diagnosis is to use disposable guided sheath (including biopsy forceps and cell brushes) which have some limitations, such as big physical damage, small biopsy tissue, etc. Cryobiospy is a new technique for biopsy developed in recent years which has many advantages over conventional biopsy, such as larger tissue, higher diagnosis yield, less complication, etc. The investigators will explore the efficacy and safety of cryobiospy vs. biopsy forceps in GGO diagnosis. The study is designed as a prospective, randomized controlled trial, 184 patients will be expected to enroll in the study and receive EBUS examination before biopsy to check whether the GGO lesions exist or not. This is a parallel-control study that patients with GGO lesions will be randomized to either TBCB group or TBFB group for biopsy. The primary aim is to compare the diagnostic yields of the two biopsy techniques. The secondary endpoint is to assess the tissue size, sampling time, number of sampling and the quality of specimen.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female aged between 18 and 80.
2. CT or other imaging examination suggest a tendency towards malignant GGO (size ≥ 8 mm). The ground glass composition is more than 50%.
3. Thin-slice CT scan with bronchial access or adjacent lesions.
4. Multidisciplinary assessment suggest that bronchopulmonary biopsy is needed to identify the pathological features of GGO.
5. It is suitable for pathological biopsy by transbronchial cryobiopsy or forceps biopsy.
6. Ability to read, understand and sign ICF.

Exclusion Criteria:

1. Disseminated GGO, suspected of benign or infectious lesions.
2. Preoperative imaging examination showed that the biopsy lesion was adjacent to the middle or large vessels.
3. There are contraindications for bronchoscopy, such as irreparable coagulation dysfunction, severe cardiopulmonary insufficiency.
4. Intolerance or difficulty in cooperating with bronchoscopy, etc.
5. Routine bronchoscopic abnormalities, such as endoscopic lesions, external pressure, mucosal lesions, stenosis, hemorrhage, etc.
6. Vulnerable groups, such as pregnant women, etc.
7. Some other special situations investigator consider subjects are not suitable to participant in this study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 184 (Estimated)
Dates: Start 2021-03-01 (Estimated); Primary Completion 2021-09-30 (Estimated); Study Completion 2021-12-30 (Estimated)

PRIMARY OUTCOMES:
Diagnostic yield | Up to 6 Months
  Diagnostic yield of transbronchial cryobiopsy (TBCB) or transbronchial forceps biopsy (TBFB) for lung ground-glass opacity.

SECONDARY OUTCOMES:
Tissue size | Up to 1 months
  The maximum diameter measured by the biopsy tissue.

OTHER OUTCOMES:
Sampling time | Up to 1 months
  The time spent in sampling the lesions begins with the insertion of biopsy tools into the bronchoscope work channel, and ends with the insertion of all biopsy specimens for the target lesion into the specimen bottle.
Number of sampling and effective sampling | Up to 1 months
  The operation for biopsy purposes is taken as one sampling, whether the sample is obtained or not, and if the sample is obtained, record as effective sampling.
Quality of specimens | Up to 6 months
  On the premise that other sample processing processes are fixed, different sampling methods will have different effects on the samples. To obtain abnormal lung tissues as eligible samples, the integrity of tissue morphology and structure preservation is an important factor in evaluating the quality of tissue samples.
Adverse events | Up to 1 months
  To evaluate the bleeding in the biopsy site mainly, which is one of the main complications of bronchoscopy biopsy. Adverse events shall be judged in accordance with relevant regulations, and serious adverse events shall be recorded and reported in accordance with regulations.

CONTACTS AND LOCATIONS:
Overall Officials: Jiayuan Sun, MD, PhD, Study Director — Shanghai Chest Hospital
Locations (1):
- Shanghai Chest Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Heidinger BH, Anderson KR, Nemec U, Costa DB, Gangadharan SP, VanderLaan PA, Bankier AA. Lung Adenocarcinoma Manifesting as Pure Ground-Glass Nodules: Correlating CT Size, Volume, Density, and Roundness with Histopathologic Invasion and Size. J Thorac Oncol. 2017 Aug;12(8):1288-1298. doi: 10.1016/j.jtho.2017.05.017. Epub 2017 May 30. PMID 28576745
- [Background] Ussavarungsi K, Kern RM, Roden AC, Ryu JH, Edell ES. Transbronchial Cryobiopsy in Diffuse Parenchymal Lung Disease: Retrospective Analysis of 74 Cases. Chest. 2017 Feb;151(2):400-408. doi: 10.1016/j.chest.2016.09.002. Epub 2016 Sep 19. PMID 27660154
- [Background] Schuhmann M, Bostanci K, Bugalho A, Warth A, Schnabel PA, Herth FJ, Eberhardt R. Endobronchial ultrasound-guided cryobiopsies in peripheral pulmonary lesions: a feasibility study. Eur Respir J. 2014 Jan;43(1):233-9. doi: 10.1183/09031936.00011313. Epub 2013 Jul 30. PMID 23900983
- [Background] Imabayashi T, Uchino J, Yoshimura A, Chihara Y, Tamiya N, Kaneko Y, Yamada T, Takayama K. Safety and Usefulness of Cryobiopsy and Stamp Cytology for the Diagnosis of Peripheral Pulmonary Lesions. Cancers (Basel). 2019 Mar 22;11(3):410. doi: 10.3390/cancers11030410. PMID 30909479
- [Background] Jiang S, Liu X, Chen J, Ma H, Xie F, Sun J. A pilot study of the ultrathin cryoprobe in the diagnosis of peripheral pulmonary ground-glass opacity lesions. Transl Lung Cancer Res. 2020 Oct;9(5):1963-1973. doi: 10.21037/tlcr-20-957. PMID 33209616
- [Background] Izumo T, Sasada S, Chavez C, Tsuchida T. The diagnostic utility of endobronchial ultrasonography with a guide sheath and tomosynthesis images for ground glass opacity pulmonary lesions. J Thorac Dis. 2013 Dec;5(6):745-50. doi: 10.3978/j.issn.2072-1439.2013.11.30. PMID 24409350
- [Background] Ikezawa Y, Sukoh N, Shinagawa N, Nakano K, Oizumi S, Nishimura M. Endobronchial ultrasonography with a guide sheath for pure or mixed ground-glass opacity lesions. Respiration. 2014;88(2):137-43. doi: 10.1159/000362885. Epub 2014 Jul 2. PMID 24993187